CLINICAL TRIAL: NCT05396014
Title: The BEST Trial: Biomarkers for Evaluating Spine Treatments
Acronym: BEST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 21-1972; 1U24AR076730 (NIH)
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2024-08

CONDITIONS: Chronic Low-back Pain
Keywords: Pain; Back Pain
MeSH Terms: conditions — Pain; Back Pain | interventions — Acceptance and Commitment Therapy; Musculoskeletal Manipulations; Duloxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Sequential Multiple Assignment Randomized Trial (SMART)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Treatment Period 1: Enhanced Self-Care (ESC) (Active Comparator): This arm includes participants who are randomized to ESC in Treatment Period 1.
  Depending on their response to Treatment 1 measured at 12 Weeks post-initial randomization, participants in this arm will stay on ESC or be randomized to augment ESC with an additional treatment during Treatment Period 2.
  Interventions: Behavioral: Enhanced Self-Care (ESC)
- Treatment Period 1: Acceptance and Commitment Therapy (ACT) (Active Comparator): This arm includes participants who are randomized to ACT in Treatment Period 1.
  Depending on their response to Treatment 1 measured at 12 Weeks post-initial randomization, participants in this arm will stay on ACT, augment ACT with an additional treatment, or switch to a new treatment during Treatment Period 2.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)
- Treatment Period 1: Evidence-Based Exercise and Manual Therapy (EBEM) (Active Comparator): This arm includes participants who are randomized to EBEM in Treatment Period 1.
  Depending on their response to Treatment 1 measured at 12 Weeks post-initial randomization, participants in this arm will stay on EBEM, augment EBEM with an additional treatment, or switch to a new treatment during Treatment Period 2.
  Interventions: Behavioral: Evidence-Based Exercise and Manual Therapy (EBEM)
- Treatment Period 1: Duloxetine (Active Comparator): This arm includes participants who are randomized to Duloxetine in Treatment Period 1.
  Depending on their response to Treatment 1 measured at 12 Weeks post-initial randomization, participants in this arm will stay on Duloxetine, augment Duloxetine with an additional treatment, or switch to a new treatment during Treatment Period 2.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Behavioral: Enhanced Self-Care (ESC) — The Enhanced Self-Care intervention will be comprised of educational modules on evidence-based cognitive-behavioral self-management skills for pain. These modules will be provided digitally for self-administration over a period of 12 weeks. There will be no therapist associated with the delivery of these educational materials; however, after the first four modules, email or text messages will be used to make personalized recommendations for accessing additional modules based upon identified problems from the baseline assessment. Additionally, the walking program module will utilize Fitbit step tracking to allow participants to monitor their walking progress.
  Arms: Treatment Period 1: Enhanced Self-Care (ESC)
Behavioral: Acceptance and Commitment Therapy (ACT) — ACT is a form of cognitive behavioral therapy that is well established for the treatment of chronic pain. The goal of ACT is to build psychological flexibility thereby interrupting pain avoidance behavior patterns. Participants randomized to ACT will take part in 12 sessions over the course of 12 weeks. Sessions will be delivered as a combination of 4 remote face-to-face visits with a therapist and 8 therapist-supported online sessions (self-directed online modules supported by provider coaching). Online sessions will focus on helping participants accept pain, connect with negative thoughts and emotions, develop mindfulness and identify and commit to values and goals that are important to them. During face-to-face sessions with the therapist, participants will be encouraged to share their experience of skills practice and mastery, provide examples of skill use at home, and describe what barriers they encountered.
  Arms: Treatment Period 1: Acceptance and Commitment Therapy (ACT)
Behavioral: Evidence-Based Exercise and Manual Therapy (EBEM) — Licensed physical therapists (PTs) or Doctors of Chiropractic (DCs) will rely on evidence-based guidance to direct decision-making on the particular type of manual and exercise therapy that may be best suited to an individual study participant. Special attention will be paid to the clinician's choice of language in regard to the purpose and expected outcomes of manual therapy in order to avoid enhancing catastrophizing ideations or preference for passive interventions. A total of 10 sessions will be provided over an 8-week treatment period. Two sessions per week are provided in the first two weeks followed by weekly sessions over the next 6 weeks. Treatment sessions will last approximately 60 minutes each.
  Arms: Treatment Period 1: Evidence-Based Exercise and Manual Therapy (EBEM)
Drug: Duloxetine — Duloxetine is a serotonin norepinephrine reuptake inhibitor (SNRI) that is FDA-approved for use in Chronic Low-Back Pain, and, as such, is included as a recommended therapy in nearly all current treatment guidelines for low back pain. Study participants will be treated with duloxetine for 12 weeks during the active treatment phase. At the time of randomization, the approved drug pharmacy at each study site will dispense between 185 and 192 duloxetine 30 mg capsules and provide to participants. This will ensure enough capsules to maintain up to a 60 mg dosage through the 12-week intervention phase and to taper the dose in the 13th week if needed.
  Other Names: Cymbalta
  Arms: Treatment Period 1: Duloxetine

SUMMARY:
The BEST Trial (Biomarkers for Evaluating Spine Treatments) is a National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)-sponsored clinical trial being conducted through the NIH Helping to End Addiction Long-term (HEAL) Initiative's Back Pain Consortium (BACPAC) Research Program. The primary objective of this trial is to inform a precision medicine approach to the treatment of Chronic Low-Back Pain by estimating the optimal treatment or combination of treatments based on patient features and response to the initial treatment. Interventions being evaluated in this trial are: (1) enhanced self-care (ESC), (2) acceptance and commitment therapy (ACT), (3) evidence-based exercise and manual therapy (EBEM), and (4) duloxetine.

DETAILED DESCRIPTION:
Each participant will complete an initial screening call and enrollment visit, followed by a 2-week run-in period, two consecutive 12-week treatment periods, and a 12-week post-treatment follow-up period. Upon completion of the run-in period, participant eligibility will be reassessed based on adherence to study protocol. Participants who no longer meet eligibility criteria will be considered screen failures and discontinued from the study.

All participants will undergo phenotyping assessments at Visit 0, 1 and 2 corresponding to baseline, the end of the first 12-week intervention period, and the end of the second 12-week intervention period, respectively. A subset of participants will undergo additional phenotyping, consisting of a more comprehensive set of phenotyping assessments, at the same visits.

Pain, Enjoyment of Life, and General Activity (PEG) and Patient Global Impressions Scale (PGIC) will be assessed at 6 weeks (midpoint of intervention period one), 12 weeks (Visit 1), 18 weeks (midpoint of intervention period two), 24 weeks (Visit 2), and 36 weeks post-baseline (12 weeks after intervention period two). Basic safety assessments will also be performed at these time points to assess participant tolerability to their current study intervention(s). Patients who are unable to tolerate their assigned study treatment will be educated on how to safely discontinue their current treatment plan but will otherwise remain in the study.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, an individual must meet all of the following inclusion criteria:

* Ability to read and understand English
* Provision of signed and dated informed consent form(s)
* Willing and able to receive study-related messages and survey links via email
* Willing and able to receive study-related phone calls
* Age 18 years old or older
* Low-back pain for at least 3 months and occurring on at least half the days in the past 6 months
* Contraindicated to no more than one of the study interventions at the time of eligibility assessment(s)
* Eligible to receive at least three of the four study interventions and willing to receive any intervention for which they are eligible
* A PEG score 4 or higher prior to the Run-in period
* Willing and able to undergo required phenotyping
* Regular reliable access to an internet-enabled device such as a smart phone, tablet, or laptop computer
* Meet Run-in period engagement eligibility criteria:

  o Completion of two Run-in study information modules prior to period 1 randomization (Visit 0)
* Low-back pain more severe than pain in other parts of the body
* Available to complete the full study protocol (approximately 9 months)

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Pregnant at the time of Visit 0 (Baseline)
* Affirmative participant response to any of the following conditions:

  * Progressive neurodegenerative disease
  * History of discitis osteomyelitis (spine infection) or spine tumor
  * History of ankylosing spondylitis, rheumatoid arthritis, polymyalgia rheumatica, psoriatic arthritis, or lupus
  * History of cauda equina syndrome or spinal radiculopathy with functional motor deficit (strength <4/5 on manual motor testing)
  * Diagnosis of any vertebral fracture in the last 6 months
  * Osteoporosis requiring pharmacologic treatment other than vitamin D, calcium supplements, or bisphosphonates.
  * History of any bone-related cancer or cancer that metastasized to the bone
  * Currently in treatment for any non-skin cancer or plan to start non-skin cancer treatment in the next 12 months
  * History of any non-skin cancer treatment in the last 24 months
  * Visual or hearing difficulties that would preclude participation
  * Uncontrolled drug/alcohol addiction
  * Individuals actively pursuing disability or workers compensation or involved in active personal injury-related litigation
  * Currently participating in another interventional pain study
* Any condition that, in the opinion of the investigator, would preclude the patient from being able to safely participate in in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1014 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Anstrom, PhD, Principal Investigator — UNC Chapel Hill; Matthew Mauck, PhD, Principal Investigator — UNC Chapel Hill; Gwendolyn Sowa, PhD, Principal Investigator — University of Pittsburgh; Daniel Clauw, MD, Principal Investigator — University of Michigan
Locations (12):
- United States (12):
  - Stanford University, Redwood City, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of Kansas Health System, Kansas City, Kansas
  - Massachusetts General Hospital/Brigham Women's Hospital, Harvard Medical School, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of North Carolina Hospital Pain Management Clinic, Chapel Hill, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
All relevant study data will be shared through NIH portals as required.
Time Frame: Data will be made publicly available on the NIH HEAL Platform or other NIH repositories after acceptance of publication for the primary results per NIH HEAL Data Sharing Policy and will remain available for a minimum of 10 years.
Access Criteria: BACPAC Data Access and Publications Policy:
  https://sites.cscc.unc.edu/cscc/sites/default/files/bacpac/qxq/BACPAC_Data_Access_and_Publications_Policy.pdf
  Data from this study may be requested by other researchers by using the HEAL Data Platform: https://heal.nih.gov/data/heal-data-ecosystem
URL: https://heal.nih.gov/data/public-access-data

REFERENCES:
- [Derived] Rowland B, Barth KS, Bell KM, Brooks AK, Chadwick AL, Cleven A, Hurley RW, Mackey S, Patel KV, Piva SR, Schneider MJ, Al-Kadhi F, Asante-Nketiah B, Bagaason S, Batorsky A, Borckardt JJ, Bowden AE, Carey TS, Castellanos J, Chen L, Chidgey B, Dalton D, Dufour JS, Eberting JL, Eller SM, Fields AJ, Fritz JM, Fu A, Ghulamhussain I, Goolsby RW, Greco CM, Grim S, Gunn CA, Hanes L, Harris RE, Harte SE, Hassett AL, Helton K, Hoffmeyer A, Ivanova A, Jones Berkeley S, Kaplan C, Kidwell KM, Knapik GG, Kosorok MR, Kurillo G, Li D, Lobo R, Long J, Lotz JC, Mageswaran P, Majumdar S, Mao J, Marras WS, McCracken LM, McCumber M, McLean SA, McMillan M, Mehling W, Mendoza R, Mitchell UH, Napadow V, O'Neill C, Pearson S, Peltier S, Rundell SD, Ryser S, Schrepf A, Schulze E, Sperger J, Vo N, Wallace MS, Wampler AM, Wasan AD, Weaver TE, Weber KA 2nd, Wilcox L, Williams DA, Wilson L, Woo JE, Zeidan F, Zhao B, Zhou B, Anstrom KJ, Clauw DJ, Sowa GA, Mauck MC. Baseline characteristics of participants in the Biomarkers for Evaluating Spine Treatments clinical trial: a sequential multiple assignment randomized trial for chronic low back paindagger. Pain Med. 2025 Nov 1;26(11):758-772. doi: 10.1093/pm/pnaf073. PMID 40794568
- [Derived] Jones Berkeley S, Wedin S, Patidar SM, Margolies SO, Goetzinger AM, Mauck MC, Wasan AD, McCracken LM. Design and implementation of online acceptance and commitment therapy with enhanced therapist support for chronic low back pain (ACT for PAIN). Pain Med. 2025 Aug 1;26(8):451-458. doi: 10.1093/pm/pnaf026. PMID 40249098
- [Derived] Mauck MC, Barth KS, Bell KM, Brooks AK, Chadwick AL, Gunn CA, Hurley RW, Ivanova A, Piva SR, Schneider MJ, Bailey JF, Bagaason S, Batorsky A, Borckardt JJ, Bowden AE, Carey TS, Castellanos J, Chen L, Chidgey B, Dalton D, Dufour JS, Fields AJ, Fritz JM, Goolsby RW, Greco CM, Harris RE, Harte S, Hassett AL, Hoffmeyer A, Jones Berkeley S, Kaplan C, Kidwell KM, Knapik GG, Kosorok MR, Kurillo G, Lobo R, Lotz JC, Mackey S, Mageswaran P, Majumdar S, Mao J, Marras WS, McCumber M, McLean SA, Mehling W, Mitchell UH, Napadow VJ, O'Neill C, Patel KV, Peltier S, Psioda M, Rowland B, Rundell SD, Schrepf A, Sperger J, Vo N, Wallace MS, Wasan AD, Weaver TE, Weber KA 2nd, Williams DA, Wilson L, Zeidan F, Zhao B, Anstrom KJ, Clauw DJ, Sowa GA. The design and rationale of the Biomarkers for Evaluating Spine Treatments trial: a sequential multiple assignment randomized trial. Pain Med. 2025 Sep 1;26(9):538-553. doi: 10.1093/pm/pnaf032. PMID 40205455

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While 1014 participants in total were enrolled in the trial, 805 were randomized. This was due to participant withdrawal or participant ineligibility during the run-in period between the enrollment visit and randomization.
Groups:
- Acceptance and Commitment Therapy (ACT) Alone: This arm included both participants who had a strong response to Acceptance and Commitment Therapy (ACT) in Period 1 and participants who were not assessed for response at the end of Period 1. In Period 1, participants randomized to ACT took part in 12 therapy sessions over the course of 12 weeks. Each participant was scheduled for a combination of 4 remote face-to-face visits and 8 therapist-supported online sessions, which included a self-directed module combined with personalized provider coaching delivered via an online messaging system. In Period 2, strong responders were encouraged to continue to practice ACT skills at home without therapist supervision and were given access to an additional 11 ACT audio modules.
- ACT Plus Duloxetine, Moderate Treatment Response: This arm included participants who had a moderate response to ACT in Period 1 and started Duloxetine in Period 2 while continuing ACT treatment.
- ACT Plus Evidence Based Exercise and Manual Therapy (EBEM), Moderate Period 1 Treatment Response: This arm included participants who had a moderate response to ACT in Period 1 and started Evidence Based Exercise and Manual Therapy (EBEM) treatment in Period 2 while continuing ACT.
- ACT Plus Enhanced Self-Care Therapy (ESC), Moderate Period 1 Treatment Response: This arm included participants who had a moderate response to ACT in Period 1 and started Enhanced Self-Care Therapy (ESC) treatment in Period 2 while continuing ACT.
- ACT Plus Duloxetine, Low Period 1 Treatment Response: This arm included participants who had a low response to ACT in Period 1 and started Duloxetine treatment in Period 2 while continuing ACT.
- ACT Plus Evidence Based Exercise and Manual Therapy (EBEM), Low Period 1 Treatment Response: This arm included participants who had a low response to ACT in Period 1 and started EBEM treatment in Period 2 while continuing ACT.
- ACT Plus Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response: This arm included participants who had a low response to ACT in Period 1 and started ESC treatment in Period 2 while continuing ACT.
- ACT Followed by Duloxetine, Low Period 1 Treatment Response: This arm included participants who had a low response to ACT in Period 1 and started Duloxetine treatment in Period 2. ACT treatment was discontinued.
- ACT Followed by Evidence Based Exercise and Manual Therapy (EBEM), Low Period 1 Treatment Response: This arm included participants who had a low response to ACT in Period 1 and started EBEM treatment in Period 2. ACT treatment was discontinued.
- ACT Followed by Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response: This arm included participants who had a low response to ACT in Period 1 and started ESC treatment in Period 2. ACT treatment was discontinued.
- ACT Followed by Duloxetine, Poor Period 1 Treatment Response: This arm included participants who had a poor response to ACT in Period 1 and started Duloxetine treatment in Period 2. ACT treatment was discontinued.
- ACT Followed by Evidence Based Exercise and Manual Therapy (EBEM), Poor Period 1 Treatment Response: This arm included participants who had a poor response to ACT in Period 1 and started EBEM treatment in Period 2. ACT treatment was discontinued.
- ACT Followed by Enhanced Self-Care Therapy (ESC), Poor Period 1 Treatment Response: This arm included participants who had a poor response to ACT in Period 1 and started ESC treatment in Period 2. ACT treatment was discontinued.
- Duloxetine Alone: This arm included both participants who had a strong response to Duloxetine in Period 1 and participants who were not assessed for response at the end of Period 1.
- Duloxetine Plus Acceptance and Commitment Therapy (ACT), Moderate Period 1 Treatment Response: This arm included participants who had a moderate response to Duloxetine in Period 1 and started ACT treatment in Period 2 while continuing Duloxetine.
- Duloxetine Plus Evidence Based Exercise & Manual Therapy(EBEM), Moderate Period 1 Treatment Response: This arm included participants who had a moderate response to Duloxetine in Period 1 and started EBEM treatment in Period 2 while continuing Duloxetine.
- Duloxetine Plus Enhanced Self-Care Therapy (ESC), Moderate Period 1 Treatment Response: This arm included participants who had a moderate response to Duloxetine in Period 1 and started ESC treatment in Period 2 while continuing Duloxetine.
- Duloxetine Plus Acceptance and Commitment Therapy (ACT), Low Period 1 Treatment Response: This arm included participants who had a low response to Duloxetine in Period 1 and started ACT treatment in Period 2 while continuing Duloxetine.
- Duloxetine Plus Evidence Based Exercise and Manual Therapy (EBEM), Low Period 1 Treatment Response: This arm included participants who had a low response to Duloxetine in Period 1 and started EBEM treatment in Period 2 while continuing Duloxetine.
- Duloxetine Plus Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response: This arm included participants who had a low response to Duloxetine in Period 1 and started ESC treatment in Period 2 while continuing Duloxetine.
- Duloxetine Followed by Acceptance and Commitment Therapy (ACT), Low Period 1 Treatment Response: This arm included participants who had a low response to Duloxetine in Period 1 and started ACT treatment in Period 2. Duloxetine treatment was discontinued.
- Duloxetine Followed by Evidence Based Exercise and Manual Therapy(EBEM), Low Period 1 Trt Response: This arm included participants who had a low response to Duloxetine in Period 1 and started EBEM treatment in Period 2. Duloxetine treatment was discontinued.
- Duloxetine Followed by Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response: This arm included participants who had a low response to Duloxetine in Period 1 and started ESC treatment in Period 2. Duloxetine treatment was discontinued.
- Duloxetine Followed by Acceptance and Commitment Therapy (ACT), Poor Period 1 Treatment Response: This arm included participants who had a poor response to Duloxetine in Period 1 and started ACT treatment in Period 2. Duloxetine treatment was discontinued.
- Duloxetine Followed by Evidence Based Exercise and Manual Therapy (EBEM), Poor Period 1 Trt Response: This arm included participants who had a poor response to Duloxetine in Period 1 and started EBEM treatment in Period 2. Duloxetine treatment was discontinued.
- Duloxetine Followed by Enhanced Self-Care Therapy (ESC), Poor Period 1 Treatment Response: This arm included participants who had a poor response to Duloxetine in Period 1 and started ESC treatment in Period 2. Duloxetine treatment was discontinued.
- Evidence Based Exercise and Manual Therapy (EBEM) Alone: This arm included both participants who had a strong response to EBEM in Period 1 and participants who were not assessed for response at the end of Period 1.
- EBEM Plus Duloxetine, Moderate Period 1 Treatment Response: This arm included participants who had a moderate response to EBEM in Period 1 and started Duloxetine treatment in Period 2 while continuing EBEM.
- EBEM Plus Acceptance and Commitment Therapy (ACT), Moderate Period 1 Treatment Response: This arm included participants who had a moderate response to EBEM in Period 1 and started ACT treatment in Period 2 while continuing EBEM.
- EBEM Plus Enhanced Self-Care Therapy (ESC), Moderate Period 1 Treatment Response: This arm included participants who had a moderate response to EBEM in Period 1 and started ESC treatment in Period 2 while continuing EBEM.
- EBEM Plus Duloxetine, Low Period 1 Treatment Response: This arm included participants who had a low response to EBEM in Period 1 and started Duloxetine treatment in Period 2 while continuing EBEM.
- EBEM Plus Acceptance and Commitment Therapy (ACT), Low Period 1 Treatment Response: This arm included participants who had a low response to EBEM in Period 1 and started ACT treatment in Period 2 while continuing EBEM.
- EBEM Plus Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response: This arm included participants who had a low response to EBEM in Period 1 and started ESC treatment in Period 2 while continuing EBEM.
- EBEM Followed by Duloxetine, Low Period 1 Treatment Response: This arm included participants who had a low response to EBEM in Period 1 and started Duloxetine treatment in Period 2. EBEM treatment was discontinued.
- EBEM Followed by Acceptance and Commitment Therapy (ACT), Low Period 1 Treatment Response: This arm included participants who had a low response to EBEM in Period 1 and started ACT treatment in Period 2. EBEM treatment was discontinued.
- EBEM Followed by Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response: This arm included participants who had a low response to ESC in Period 1 and started Duloxetine treatment in Period 2. EBEM treatment was discontinued.
- EBEM Followed by Duloxetine, Poor Period 1 Treatment Response: This arm included participants who had a poor response to EBEM in Period 1 and started Duloxetine treatment in Period 2. EBEM treatment was discontinued.
- EBEM Followed by Acceptance and Commitment Therapy (ACT), Poor Period 1 Treatment Response: This arm included participants who had a poor response to EBEM in Period 1 and started ACT treatment in Period 2. EBEM treatment was discontinued.
- EBEM Followed by Enhanced Self-Care Therapy (ESC), Poor Period 1 Treatment Response: This arm included participants who had a poor response to EBEM in Period 1 and started ESC treatment in Period 2. EBEM treatment was discontinued.
- Enhanced Self-Care Therapy (ESC) Alone: This arm included both participants who had a strong response to ESC in Period 1 and participants who were not assessed for response at the end of Period 1.
- ESC Plus Duloxetine, Moderate to Low Period 1 Treatment Response: This arm included participants who had a moderate to poor response to ESC in Period 1 and started Duloxetine treatment in Period 2. ESC treatment was discontinued.
- ESC Plus Acceptance and Commitment Therapy (ACT), Moderate to Low Period 1 Treatment Response: This arm included participants who had a moderate to poor response to ESC in Period 1 and started ACT treatment in Period 2. ESC treatment was discontinued.
- ESC Plus Evidence Based Exercise and Manual Therapy (EBEM), Moderate to Low Period 1 Trt Response: This arm included participants who had a moderate to poor response to ESC in Period 1 and started EBEM treatment in Period 2. ESC treatment was discontinued.
Period: Stage 1 Intervention (Weeks 0-12)
Arm/Group | Acceptance and Commitment Therapy (ACT) Alone | ACT Plus Duloxetine, Moderate Treatment Response | ACT Plus Evidence Based Exercise and Manual Therapy (EBEM), Moderate Period 1 Treatment Response | ACT Plus Enhanced Self-Care Therapy (ESC), Moderate Period 1 Treatment Response | ACT Plus Duloxetine, Low Period 1 Treatment Response | ACT Plus Evidence Based Exercise and Manual Therapy (EBEM), Low Period 1 Treatment Response | ACT Plus Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response | ACT Followed by Duloxetine, Low Period 1 Treatment Response | ACT Followed by Evidence Based Exercise and Manual Therapy (EBEM), Low Period 1 Treatment Response | ACT Followed by Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response | ACT Followed by Duloxetine, Poor Period 1 Treatment Response | ACT Followed by Evidence Based Exercise and Manual Therapy (EBEM), Poor Period 1 Treatment Response | ACT Followed by Enhanced Self-Care Therapy (ESC), Poor Period 1 Treatment Response | Duloxetine Alone | Duloxetine Plus Acceptance and Commitment Therapy (ACT), Moderate Period 1 Treatment Response | Duloxetine Plus Evidence Based Exercise & Manual Therapy(EBEM), Moderate Period 1 Treatment Response | Duloxetine Plus Enhanced Self-Care Therapy (ESC), Moderate Period 1 Treatment Response | Duloxetine Plus Acceptance and Commitment Therapy (ACT), Low Period 1 Treatment Response | Duloxetine Plus Evidence Based Exercise and Manual Therapy (EBEM), Low Period 1 Treatment Response | Duloxetine Plus Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response | Duloxetine Followed by Acceptance and Commitment Therapy (ACT), Low Period 1 Treatment Response | Duloxetine Followed by Evidence Based Exercise and Manual Therapy(EBEM), Low Period 1 Trt Response | Duloxetine Followed by Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response | Duloxetine Followed by Acceptance and Commitment Therapy (ACT), Poor Period 1 Treatment Response | Duloxetine Followed by Evidence Based Exercise and Manual Therapy (EBEM), Poor Period 1 Trt Response | Duloxetine Followed by Enhanced Self-Care Therapy (ESC), Poor Period 1 Treatment Response | Evidence Based Exercise and Manual Therapy (EBEM) Alone | EBEM Plus Duloxetine, Moderate Period 1 Treatment Response | EBEM Plus Acceptance and Commitment Therapy (ACT), Moderate Period 1 Treatment Response | EBEM Plus Enhanced Self-Care Therapy (ESC), Moderate Period 1 Treatment Response | EBEM Plus Duloxetine, Low Period 1 Treatment Response | EBEM Plus Acceptance and Commitment Therapy (ACT), Low Period 1 Treatment Response | EBEM Plus Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response | EBEM Followed by Duloxetine, Low Period 1 Treatment Response | EBEM Followed by Acceptance and Commitment Therapy (ACT), Low Period 1 Treatment Response | EBEM Followed by Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response | EBEM Followed by Duloxetine, Poor Period 1 Treatment Response | EBEM Followed by Acceptance and Commitment Therapy (ACT), Poor Period 1 Treatment Response | EBEM Followed by Enhanced Self-Care Therapy (ESC), Poor Period 1 Treatment Response | Enhanced Self-Care Therapy (ESC) Alone | ESC Plus Duloxetine, Moderate to Low Period 1 Treatment Response | ESC Plus Acceptance and Commitment Therapy (ACT), Moderate to Low Period 1 Treatment Response | ESC Plus Evidence Based Exercise and Manual Therapy (EBEM), Moderate to Low Period 1 Trt Response
Started | 63 | 8 | 8 | 5 | 12 | 21 | 20 | 12 | 22 | 28 | 2 | 1 | 1 | 71 | 9 | 4 | 4 | 4 | 8 | 9 | 25 | 26 | 26 | 4 | 3 | 5 | 97 | 5 | 15 | 12 | 6 | 9 | 14 | 13 | 12 | 7 | 4 | 1 | 4 | 46 | 41 | 59 | 59
Completed | 28 | 8 | 8 | 5 | 12 | 21 | 20 | 12 | 22 | 28 | 2 | 1 | 1 | 48 | 9 | 4 | 4 | 4 | 8 | 9 | 25 | 26 | 26 | 4 | 3 | 5 | 71 | 5 | 15 | 12 | 6 | 9 | 14 | 13 | 12 | 7 | 4 | 1 | 4 | 16 | 41 | 59 | 59
Not Completed | 35 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 30 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 0 | 0 | 0
Not completed — Lost to Follow-up | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2 Screening (Week 12 Pre-Rand.)
Arm/Group | Acceptance and Commitment Therapy (ACT) Alone | ACT Plus Duloxetine, Moderate Treatment Response | ACT Plus Evidence Based Exercise and Manual Therapy (EBEM), Moderate Period 1 Treatment Response | ACT Plus Enhanced Self-Care Therapy (ESC), Moderate Period 1 Treatment Response | ACT Plus Duloxetine, Low Period 1 Treatment Response | ACT Plus Evidence Based Exercise and Manual Therapy (EBEM), Low Period 1 Treatment Response | ACT Plus Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response | ACT Followed by Duloxetine, Low Period 1 Treatment Response | ACT Followed by Evidence Based Exercise and Manual Therapy (EBEM), Low Period 1 Treatment Response | ACT Followed by Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response | ACT Followed by Duloxetine, Poor Period 1 Treatment Response | ACT Followed by Evidence Based Exercise and Manual Therapy (EBEM), Poor Period 1 Treatment Response | ACT Followed by Enhanced Self-Care Therapy (ESC), Poor Period 1 Treatment Response | Duloxetine Alone | Duloxetine Plus Acceptance and Commitment Therapy (ACT), Moderate Period 1 Treatment Response | Duloxetine Plus Evidence Based Exercise & Manual Therapy(EBEM), Moderate Period 1 Treatment Response | Duloxetine Plus Enhanced Self-Care Therapy (ESC), Moderate Period 1 Treatment Response | Duloxetine Plus Acceptance and Commitment Therapy (ACT), Low Period 1 Treatment Response | Duloxetine Plus Evidence Based Exercise and Manual Therapy (EBEM), Low Period 1 Treatment Response | Duloxetine Plus Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response | Duloxetine Followed by Acceptance and Commitment Therapy (ACT), Low Period 1 Treatment Response | Duloxetine Followed by Evidence Based Exercise and Manual Therapy(EBEM), Low Period 1 Trt Response | Duloxetine Followed by Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response | Duloxetine Followed by Acceptance and Commitment Therapy (ACT), Poor Period 1 Treatment Response | Duloxetine Followed by Evidence Based Exercise and Manual Therapy (EBEM), Poor Period 1 Trt Response | Duloxetine Followed by Enhanced Self-Care Therapy (ESC), Poor Period 1 Treatment Response | Evidence Based Exercise and Manual Therapy (EBEM) Alone | EBEM Plus Duloxetine, Moderate Period 1 Treatment Response | EBEM Plus Acceptance and Commitment Therapy (ACT), Moderate Period 1 Treatment Response | EBEM Plus Enhanced Self-Care Therapy (ESC), Moderate Period 1 Treatment Response | EBEM Plus Duloxetine, Low Period 1 Treatment Response | EBEM Plus Acceptance and Commitment Therapy (ACT), Low Period 1 Treatment Response | EBEM Plus Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response | EBEM Followed by Duloxetine, Low Period 1 Treatment Response | EBEM Followed by Acceptance and Commitment Therapy (ACT), Low Period 1 Treatment Response | EBEM Followed by Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response | EBEM Followed by Duloxetine, Poor Period 1 Treatment Response | EBEM Followed by Acceptance and Commitment Therapy (ACT), Poor Period 1 Treatment Response | EBEM Followed by Enhanced Self-Care Therapy (ESC), Poor Period 1 Treatment Response | Enhanced Self-Care Therapy (ESC) Alone | ESC Plus Duloxetine, Moderate to Low Period 1 Treatment Response | ESC Plus Acceptance and Commitment Therapy (ACT), Moderate to Low Period 1 Treatment Response | ESC Plus Evidence Based Exercise and Manual Therapy (EBEM), Moderate to Low Period 1 Trt Response
Started | 28 | 8 | 8 | 5 | 12 | 21 | 20 | 12 | 22 | 28 | 2 | 1 | 1 | 48 | 9 | 4 | 4 | 4 | 8 | 9 | 25 | 26 | 26 | 4 | 3 | 5 | 71 | 5 | 15 | 12 | 6 | 9 | 14 | 13 | 12 | 7 | 4 | 1 | 4 | 16 | 41 | 59 | 59
Completed | 26 | 8 | 8 | 5 | 12 | 21 | 20 | 12 | 22 | 28 | 2 | 1 | 1 | 45 | 9 | 4 | 4 | 4 | 8 | 9 | 25 | 26 | 26 | 4 | 3 | 5 | 70 | 5 | 15 | 12 | 6 | 9 | 14 | 13 | 12 | 7 | 4 | 1 | 4 | 14 | 41 | 59 | 59
Not Completed | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2 Intervention (Weeks 12-24)
Arm/Group | Acceptance and Commitment Therapy (ACT) Alone | ACT Plus Duloxetine, Moderate Treatment Response | ACT Plus Evidence Based Exercise and Manual Therapy (EBEM), Moderate Period 1 Treatment Response | ACT Plus Enhanced Self-Care Therapy (ESC), Moderate Period 1 Treatment Response | ACT Plus Duloxetine, Low Period 1 Treatment Response | ACT Plus Evidence Based Exercise and Manual Therapy (EBEM), Low Period 1 Treatment Response | ACT Plus Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response | ACT Followed by Duloxetine, Low Period 1 Treatment Response | ACT Followed by Evidence Based Exercise and Manual Therapy (EBEM), Low Period 1 Treatment Response | ACT Followed by Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response | ACT Followed by Duloxetine, Poor Period 1 Treatment Response | ACT Followed by Evidence Based Exercise and Manual Therapy (EBEM), Poor Period 1 Treatment Response | ACT Followed by Enhanced Self-Care Therapy (ESC), Poor Period 1 Treatment Response | Duloxetine Alone | Duloxetine Plus Acceptance and Commitment Therapy (ACT), Moderate Period 1 Treatment Response | Duloxetine Plus Evidence Based Exercise & Manual Therapy(EBEM), Moderate Period 1 Treatment Response | Duloxetine Plus Enhanced Self-Care Therapy (ESC), Moderate Period 1 Treatment Response | Duloxetine Plus Acceptance and Commitment Therapy (ACT), Low Period 1 Treatment Response | Duloxetine Plus Evidence Based Exercise and Manual Therapy (EBEM), Low Period 1 Treatment Response | Duloxetine Plus Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response | Duloxetine Followed by Acceptance and Commitment Therapy (ACT), Low Period 1 Treatment Response | Duloxetine Followed by Evidence Based Exercise and Manual Therapy(EBEM), Low Period 1 Trt Response | Duloxetine Followed by Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response | Duloxetine Followed by Acceptance and Commitment Therapy (ACT), Poor Period 1 Treatment Response | Duloxetine Followed by Evidence Based Exercise and Manual Therapy (EBEM), Poor Period 1 Trt Response | Duloxetine Followed by Enhanced Self-Care Therapy (ESC), Poor Period 1 Treatment Response | Evidence Based Exercise and Manual Therapy (EBEM) Alone | EBEM Plus Duloxetine, Moderate Period 1 Treatment Response | EBEM Plus Acceptance and Commitment Therapy (ACT), Moderate Period 1 Treatment Response | EBEM Plus Enhanced Self-Care Therapy (ESC), Moderate Period 1 Treatment Response | EBEM Plus Duloxetine, Low Period 1 Treatment Response | EBEM Plus Acceptance and Commitment Therapy (ACT), Low Period 1 Treatment Response | EBEM Plus Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response | EBEM Followed by Duloxetine, Low Period 1 Treatment Response | EBEM Followed by Acceptance and Commitment Therapy (ACT), Low Period 1 Treatment Response | EBEM Followed by Enhanced Self-Care Therapy (ESC), Low Period 1 Treatment Response | EBEM Followed by Duloxetine, Poor Period 1 Treatment Response | EBEM Followed by Acceptance and Commitment Therapy (ACT), Poor Period 1 Treatment Response | EBEM Followed by Enhanced Self-Care Therapy (ESC), Poor Period 1 Treatment Response | Enhanced Self-Care Therapy (ESC) Alone | ESC Plus Duloxetine, Moderate to Low Period 1 Treatment Response | ESC Plus Acceptance and Commitment Therapy (ACT), Moderate to Low Period 1 Treatment Response | ESC Plus Evidence Based Exercise and Manual Therapy (EBEM), Moderate to Low Period 1 Trt Response
Started | 26 | 8 | 8 | 5 | 12 | 21 | 20 | 12 | 22 | 28 | 2 | 1 | 1 | 45 | 9 | 4 | 4 | 4 | 8 | 9 | 25 | 26 | 26 | 4 | 3 | 5 | 70 | 5 | 15 | 12 | 6 | 9 | 14 | 13 | 12 | 7 | 4 | 1 | 4 | 14 | 41 | 59 | 59
Completed | 26 | 8 | 8 | 3 | 12 | 20 | 18 | 12 | 18 | 27 | 2 | 1 | 1 | 43 | 9 | 3 | 3 | 3 | 7 | 9 | 25 | 25 | 23 | 3 | 1 | 2 | 67 | 4 | 15 | 12 | 5 | 7 | 13 | 13 | 9 | 5 | 4 | 1 | 4 | 14 | 37 | 54 | 56
Not Completed | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 4 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 3 | 1 | 2 | 3 | 3 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 4 | 5 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stage 1: Acceptance and Commitment Therapy (ACT): ACT is a form of cognitive behavioral therapy that is well established for the treatment of chronic pain. The goal of ACT is to build psychological flexibility thereby interrupting pain avoidance behavior patterns. Participants randomized to ACT will take part in 12 sessions over the course of 12 weeks. Sessions will be delivered as a combination of 4 remote face-to-face visits with a therapist and 8 therapist-supported online sessions (self-directed online modules supported by provider coaching). Online sessions will focus on helping participants accept pain, connect with negative thoughts and emotions, develop mindfulness and identify and commit to values and goals that are important to them. During face-to-face sessions with the therapist, participants will be encouraged to share their experience of skills practice and mastery, provide examples of skill use at home, and describe what barriers they encountered.
- Stage 1: Duloxetine: Duloxetine is a serotonin norepinephrine reuptake inhibitor (SNRI) that is FDA-approved for use in Chronic Low-Back Pain, and, as such, is included as a recommended therapy in nearly all current treatment guidelines for low back pain. Study participants will be treated with duloxetine for 12 weeks during the active treatment phase. At the time of randomization, the approved drug pharmacy at each study site will dispense between 185 and 192 duloxetine 30 mg capsules and provide to participants. This will ensure enough capsules to maintain up to a 60 mg dosage through the 12-week intervention phase and to taper the dose in the 13th week if needed.
- Stage 1: Evidence Based Exercise and Manual Therapy (EBEM): Licensed physical therapists (PTs) or Doctors of Chiropractic (DCs) will rely on evidence-based guidance to direct decision-making on the particular type of manual and exercise therapy that may be best suited to an individual study participant. Special attention will be paid to the clinician's choice of language in regard to the purpose and expected outcomes of manual therapy in order to avoid enhancing catastrophizing ideations or preference for passive interventions. A total of 10 sessions will be provided over an 8-week treatment period. Two sessions per week are provided in the first two weeks followed by weekly sessions over the next 6 weeks. Treatment sessions will last approximately 60 minutes each.
- Stage 1: Enhanced Self-Care Therapy (ESC): The Enhanced Self-Care intervention will be comprised of educational modules on evidence-based cognitive-behavioral self-management skills for pain. These modules will be provided digitally for self-administration over a period of 12 weeks. There will be no therapist associated with the delivery of these educational materials; however, after the first four modules, email or text messages will be used to make personalized recommendations for accessing additional modules based upon identified problems from the baseline assessment. Additionally, the walking program module will utilize Fitbit step tracking to allow participants to monitor their walking progress.
- Total: Total of all reporting groups
Arm/Group | Stage 1: Acceptance and Commitment Therapy (ACT) | Stage 1: Duloxetine | Stage 1: Evidence Based Exercise and Manual Therapy (EBEM) | Stage 1: Enhanced Self-Care Therapy (ESC) | Total
Number analyzed (Participants) | 203 | 198 | 199 | 205 | 805
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 166 | 160 | 161 | 164 | 651
  >=65 years | 37 | 38 | 38 | 41 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (16.5) | 51.6 (15.4) | 49.5 (16.3) | 51.2 (16.1) | 50.4 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 115 | 131 | 134 | 496
  Male | 87 | 83 | 68 | 71 | 309
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 13 | 17 | 18 | 72
  Not Hispanic or Latino | 172 | 182 | 178 | 187 | 719
  Unknown or Not Reported | 7 | 3 | 4 | 0 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 1 | 3
  Asian | 23 | 21 | 17 | 19 | 80
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 2 | 3
  Black or African American | 21 | 19 | 21 | 29 | 90
  White | 142 | 144 | 144 | 142 | 572
  More than one race | 6 | 6 | 7 | 8 | 27
  Unknown or Not Reported | 10 | 7 | 9 | 4 | 30
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 203 | 198 | 199 | 205 | 805
Highest Level of Education Completed [Count of Participants; unit: Participants]
  Did not complete Secondary School or High School | 6 | 6 | 8 | 8 | 28
  High School or Secondary School Degree Complete | 31 | 24 | 33 | 41 | 129
  Associate's or Technical Degree Complete | 33 | 27 | 36 | 35 | 131
  College or Baccalaureate Degree Complete | 75 | 85 | 65 | 69 | 294
  Doctoral or Postgraduate Education | 56 | 56 | 57 | 51 | 220
  Missing | 2 | 0 | 0 | 1 | 3
Current Employment Status [Count of Participants; unit: Participants]
  Full-time employment | 102 | 101 | 112 | 84 | 399
  Not employed | 64 | 72 | 60 | 83 | 279
  Part-time employment | 35 | 25 | 27 | 37 | 124
  Missing | 2 | 0 | 0 | 1 | 3
Current Relationship Status [Count of Participants; unit: Participants]
  Married | 97 | 117 | 94 | 99 | 407
  Never Married | 53 | 37 | 49 | 46 | 185
  Domestic Partner | 13 | 12 | 17 | 10 | 52
  Widowed | 6 | 11 | 6 | 7 | 30
  Divorced or Separated | 32 | 21 | 33 | 42 | 128
  Missing | 2 | 0 | 0 | 1 | 3
Number of People Living in Household [Count of Participants; unit: Participants]
  1 | 50 | 43 | 53 | 58 | 204
  2 | 85 | 88 | 62 | 87 | 322
  3 | 30 | 25 | 40 | 19 | 114
  4 | 25 | 29 | 29 | 23 | 106
  5 | 8 | 9 | 8 | 13 | 38
  6 | 3 | 3 | 7 | 1 | 14
  7 | 0 | 1 | 0 | 1 | 2
  8 | 0 | 0 | 0 | 2 | 2
  Missing | 2 | 0 | 0 | 1 | 3
Annual household income from all sources [Count of Participants; unit: Participants]
  Less than $10,000 | 11 | 4 | 9 | 12 | 36
  $10,000 to $24,999 | 20 | 14 | 16 | 23 | 73
  $25,000 to $34,999 | 15 | 11 | 15 | 16 | 57
  $35,000 to $49,999 | 15 | 15 | 21 | 13 | 64
  $50,000 to $74,999 | 24 | 21 | 25 | 20 | 90
  $75,000 to $99,999 | 21 | 19 | 22 | 28 | 90
  $100,000 to $149,999 | 31 | 24 | 34 | 39 | 128
  $150,000 to $199,999 | 17 | 21 | 14 | 6 | 58
  $200,000 or more | 22 | 39 | 20 | 20 | 101
  Prefer not to answer | 0 | 0 | 0 | 0 | 0
  Missing | 27 | 30 | 23 | 28 | 108
Pain, Enjoyment of Life, General Activity (PEG) score [Mean (Standard Deviation); unit: units on a scale] — The PEG scale, a subset of the Brief Pain Inventory (BPI), evaluates pain intensity and its impact on enjoyment of life and general activity (i.e., pain interference) using a ranked scale (score 0 = "No Pain" or "Does not Interfere" to 10 = "Pain as bad as you can imagine" or "Completely Interferes"). Each component (Pain, Enjoyment of Life, and General Activity) is on a 0-10 scale, with an average score taken of the three, and with a higher average score reflecting greater disruption in daily functioning.
  units on a scale | 5.4 (2.0) | 5.1 (1.9) | 5.3 (1.8) | 5.5 (1.9) | 5.3 (1.9)
Pain, Enjoyment of Life, General Activity (PEG) score, median (range) [Median (Full Range); unit: units on a scale] — The PEG scale, a subset of the Brief Pain Inventory (BPI), evaluates pain intensity and its impact on enjoyment of life and general activity (i.e., pain interference) using a ranked scale (score 0 = "No Pain" or "Does not Interfere" to 10 = "Pain as bad as you can imagine" or "Completely Interferes"). Each component (Pain, Enjoyment of Life, and General Activity) is on a 0-10 scale, with an average score taken of the three, and with a higher average score reflecting greater disruption in daily functioning.
  units on a scale | 5.3 [0.7 to 10.0] | 5.0 [0.7 to 9.7] | 5.3 [0.7 to 10.0] | 5.3 [1.0 to 9.7] | 5.3 [0.7 to 10.0]
Self-reported low back pain duration (months) [Mean (Standard Deviation); unit: months] | 163.4 (150.0) | 156.7 (151.0) | 156.4 (139.8) | 154.7 (123.4) | 157.8 (141.2)
Self-reported low back pain duration [Count of Participants; unit: Participants]
  <1 year | 12 | 14 | 9 | 15 | 50
  1-5 years | 70 | 66 | 71 | 67 | 274
  >5 years | 121 | 118 | 119 | 123 | 481
  Missing | 0 | 0 | 0 | 0 | 0
Low Back Pain Frequency in the past 6 months [Count of Participants; unit: Participants]
  Every day or nearly every day | 181 | 163 | 160 | 169 | 673
  At least half the days | 22 | 35 | 39 | 36 | 132
Low Back Pain Specific Pain Intensity [Mean (Standard Deviation); unit: units on a scale] — Low-Back Pain Specific Pain Intensity measures pain intensity using a single, 10-point ranked scale (score 0 = "No Pain" to 10 = "Worst Imaginable Pain") where a higher score reflects greater pain intensity.
  units on a scale | 5.6 (1.9) | 5.4 (1.8) | 5.6 (1.7) | 5.8 (1.7) | 5.6 (1.8)
Low Back Pain Specific Pain Intensity, median (range) [Median (Full Range); unit: units on a scale] — Low-Back Pain Specific Pain Intensity measures pain intensity using a single, 10-point ranked scale (score 0 = "No Pain" to 10 = "Worst Imaginable Pain") where a higher score reflects greater pain intensity.
  units on a scale | 5.0 [1.0 to 10.0] | 6.0 [1.0 to 10.0] | 6.0 [1.0 to 10.0] | 6.0 [1.0 to 9.0] | 6.0 [1.0 to 10.0]
Ever had low back operation [Count of Participants; unit: Participants]
  No | 176 | 174 | 177 | 171 | 698
  Yes, at least one | 25 | 24 | 22 | 33 | 104
  Missing | 2 | 0 | 0 | 1 | 3
When was last back operation [Count of Participants; unit: Participants] — Population: The number of participants analyzed are participants who had a low back operation.
  Participants
    number analyzed (Participants) | 25 | 24 | 22 | 33 | 104
    Less than 6 months ago | 20 | 18 | 15 | 21 | 74
    More than 6 months ago but less than 1 year ago | 5 | 6 | 7 | 12 | 30
    Between 1 and 2 years ago | 0 | 0 | 0 | 0 | 0
    More than 2 years ago | 0 | 0 | 0 | 0 | 0
Any back operations involve a spinal fusion [Count of Participants; unit: Participants] — Population: The number of participants analyzed are those who had a low back operation.
  Participants
    number analyzed (Participants) | 25 | 24 | 22 | 33 | 104
    No | 15 | 13 | 13 | 20 | 61
    Yes | 7 | 9 | 7 | 10 | 33
    Not Sure | 3 | 2 | 2 | 3 | 10
Ever unemployed for 1 or more months due to low back pain [Count of Participants; unit: Participants]
  No | 145 | 151 | 142 | 134 | 572
  Yes | 40 | 27 | 36 | 43 | 146
  Does not apply | 16 | 20 | 21 | 27 | 84
  Missing | 2 | 0 | 0 | 1 | 3
Ever filed or awarded worker's compensation claim related to back problem [Count of Participants; unit: Participants]
  No | 179 | 176 | 175 | 174 | 704
  Yes | 6 | 9 | 7 | 7 | 29
  Does not apply | 16 | 13 | 17 | 23 | 69
  Missing | 2 | 0 | 0 | 1 | 3
Involved in a lawsuit or legal claim related to back problem [Count of Participants; unit: Participants]
  No | 199 | 196 | 198 | 201 | 794
  Yes | 0 | 1 | 0 | 1 | 2
  Not sure | 2 | 1 | 1 | 2 | 6
  Missing | 2 | 0 | 0 | 1 | 3
Ever applied for, or received, disability insurance for pain condition [Count of Participants; unit: Participants]
  No | 180 | 185 | 183 | 170 | 718
  Yes | 21 | 13 | 16 | 34 | 84
  Missing | 2 | 0 | 0 | 1 | 3
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.8 (6.3) | 29.3 (7.2) | 29.0 (6.3) | 29.4 (6.9) | 29.1 (6.7)
Systolic Blood Pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 125.8 (15.5) | 129.5 (17.2) | 124.2 (14.3) | 125.6 (13.6) | 126.3 (15.3)
Diastolic Blood Pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 78.5 (10.5) | 78.7 (10.2) | 76.7 (9.6) | 77.7 (10.1) | 77.9 (10.1)
Heart Rate (bpm) [Mean (Standard Deviation); unit: bpm] | 71.7 (12.9) | 70.9 (11.6) | 73.2 (12.0) | 72.8 (12.3) | 72.2 (12.2)
Ever Hip Replacement Surgery [Count of Participants; unit: Participants]
  Yes | 7 | 7 | 9 | 9 | 32
  No | 196 | 191 | 190 | 196 | 773
  Missing | 0 | 0 | 0 | 0 | 0
Ever Knee Replacement Surgery [Count of Participants; unit: Participants]
  Yes | 13 | 13 | 15 | 9 | 50
  No | 190 | 185 | 184 | 196 | 755
  Missing | 0 | 0 | 0 | 0 | 0
Observed Gait [Count of Participants; unit: Participants]
  Normal | 179 | 164 | 172 | 169 | 684
  Antalgic | 24 | 34 | 27 | 36 | 121
  Missing | 0 | 0 | 0 | 0 | 0
TAPS Tobacco Use [Count of Participants; unit: Participants] — The Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) Tool Part 1 is a 4-item screening for tobacco use, alcohol use, prescription medication misuse, and illicit substance use in the past year (i.e., previous 12 months). Each of the four multiple-choice items has five possible responses to choose from (0=Daily or Almost Daily to 4=Never). For each item, higher scores indicate better outcome.
  Participants
    Daily or Almost Daily | 14 | 15 | 14 | 25 | 68
    Less Than Daily | 18 | 17 | 17 | 20 | 72
    Never | 169 | 166 | 168 | 159 | 662
    Missing | 2 | 0 | 0 | 1 | 3
TAPS Alcohol Use [Count of Participants; unit: Participants] — The Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) Tool Part 1 is a 4-item screening for tobacco use, alcohol use, prescription medication misuse, and illicit substance use in the past year (i.e., previous 12 months). Each of the four multiple-choice items has five possible responses to choose from (0=Daily or Almost Daily to 4=Never). For each item, higher scores indicate better outcome.
  Participants
    At Least Weekly | 15 | 12 | 13 | 11 | 51
    Monthly | 8 | 15 | 12 | 25 | 60
    Less Than Monthly | 52 | 52 | 52 | 46 | 202
    Never | 125 | 118 | 122 | 122 | 487
    Missing | 3 | 1 | 0 | 1 | 5
TAPS Drug Use [Count of Participants; unit: Participants] — The Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) Tool Part 1 is a 4-item screening for tobacco use, alcohol use, prescription medication misuse, and illicit substance use in the past year (i.e., previous 12 months). Each of the four multiple-choice items has five possible responses to choose from (0=Daily or Almost Daily to 4=Never). For each item, higher scores indicate better outcome.
  Participants
    Daily or Almost Daily | 11 | 5 | 8 | 11 | 35
    Between Monthly to Weekly | 14 | 8 | 11 | 13 | 46
    Less Than Monthly | 11 | 17 | 13 | 22 | 63
    Never | 165 | 168 | 167 | 158 | 658
    Missing | 2 | 0 | 0 | 1 | 3
TAPS Prescription Drug Used Not as Intended [Count of Participants; unit: Participants] — The Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) Tool Part 1 is a 4-item screening for tobacco use, alcohol use, prescription medication misuse, and illicit substance use in the past year (i.e., previous 12 months). Each of the four multiple-choice items has five possible responses to choose from (0=Daily or Almost Daily to 4=Never). For each item, higher scores indicate better outcome.
  Participants
    At Least Once | 13 | 16 | 12 | 19 | 60
    Never | 188 | 182 | 187 | 185 | 742
    Missing | 2 | 0 | 0 | 1 | 3
Currently Taking Opioid Medication (daily) [Count of Participants; unit: Participants]
  Yes | 11 | 8 | 9 | 13 | 41
  No | 192 | 190 | 190 | 192 | 764
  Not Sure | 0 | 0 | 0 | 0 | 0
Previously Diagnosed with Coronavirus Disease 2019 (COVID-19) [Count of Participants; unit: Participants]
  Yes | 112 | 98 | 107 | 104 | 421
  No | 84 | 95 | 85 | 98 | 362
  Not Sure | 4 | 5 | 5 | 1 | 15
  Prefer not to answer | 3 | 0 | 2 | 2 | 7
  Missing | 0 | 0 | 0 | 0 | 0
Long COVID [Count of Participants; unit: Participants]
  Yes | 20 | 18 | 21 | 23 | 82
  No | 79 | 74 | 81 | 74 | 308
  Not Sure | 13 | 6 | 5 | 7 | 31
  Prefer not to answer | 0 | 0 | 0 | 0 | 0
  No self-reported COVID-19 diagnosis | 91 | 100 | 92 | 101 | 384
COVID-19 Vaccine [Count of Participants; unit: Participants]
  Yes | 186 | 188 | 182 | 189 | 745
  No | 15 | 8 | 17 | 14 | 54
  Not Sure | 0 | 0 | 0 | 0 | 0
  Prefer Not to Answer | 2 | 2 | 0 | 2 | 6
Fear-Avoidance Beliefs - Physical Activity (FABQ-PA) Score [Mean (Standard Deviation); unit: units on a scale] — The Fear-Avoidance Beliefs - Physical Activity (FABQ-PA) questionnaire consists of 4 items measuring fear-avoidance of physical activity. A patient rates their agreement with each statement on a 7-point Likert scale where 0= completely disagree and 6=completely agree. The total score is the sum of individual questions with a total score range of 0-24. Higher scores indicate a greater tendency to avoid physical activity due to fear (i.e., higher fear-avoidance).
  units on a scale | 13.7 (5.1) | 12.3 (5.4) | 13.3 (5.2) | 13.4 (5.6) | 13.2 (5.3)
Generalized Anxiety Disorder (GAD-2) Raw Score [Mean (Standard Deviation); unit: units on a scale] — GAD-2 consists of 2 items and measures how often one has been bothered by anxiety-related problems. Each is answered with a score of 0 (not at all) to 3 (nearly every day). The total score is the sum of individual questions with a total score range of 0-6; the higher the score, the more frequent one is bothered by anxiety.
  units on a scale | 1.7 (1.8) | 1.1 (1.2) | 1.5 (1.7) | 1.4 (1.6) | 1.4 (1.6)
Keele STarT Back Screening Tool Risk [Count of Participants; unit: Participants] — A 9-item questionnaire assessing physical and psychosocial factors that can contribute to persistent low back pain. The psychosocial subscale (5-items) helps differentiate between medium and high-risk groups. The first eight questions are disagree (0) or agree (1). The last question is a scale of 0 (Not at all) to 4 (Extremely). The total score ranges from 0-9 with higher scores indicating higher risk. The total raw score and subscore categorize low risk (total = 3 or less), medium risk (total = 4+ and subscore = 3 or less), and high risk (total = 4+ and subscore = 4+) groups.
  Participants
    Low Risk | 72 | 92 | 73 | 79 | 316
    Medium Risk | 100 | 79 | 80 | 86 | 345
    High Risk | 31 | 27 | 44 | 40 | 142
    Missing | 0 | 0 | 2 | 0 | 2
Oswestry Disability Index (ODI) Percentage [Mean (Standard Deviation); unit: units on a scale] — A 10-item questionnaire used to measure disability related to low back pain. Each question is scored from 0-5 (minimum to maximum). The percentage of disability is the sum all the responses, divided by the total number of questions answered multiplied by 5, then multiplied by 100 (i.e., total scored / total possible score x 100). The score ranges from 0% (no disability) to 100% (most severe disability). Scores from 0% to 20% indicate minimal disability; 20% to 40%, moderate disability; 40% to 60%, severe disability; 60% to 80%, crippled; and 80% to 100%, bedbound or exaggerating.
  units on a scale | 29.4 (13.5) | 27.7 (12.0) | 30.7 (14.1) | 31.1 (14.3) | 29.8 (13.6)
Oswestry Disability Index (ODI) Percentage, median (range) [Median (Full Range); unit: units on a scale] — A 10-item questionnaire used to measure disability related to low back pain. Each question is scored from 0-5 (minimum to maximum). The percentage of disability is the sum all the responses, divided by the total number of questions answered multiplied by 5, then multiplied by 100 (i.e., total scored / total possible score x 100). The score ranges from 0% (no disability) to 100% (most severe disability). Scores from 0% to 20% indicate minimal disability; 20% to 40%, moderate disability; 40% to 60%, severe disability; 60% to 80%, crippled; and 80% to 100%, bedbound or exaggerating.
  units on a scale | 28.0 [4.0 to 86.7] | 26.7 [4.4 to 70.0] | 28.0 [6.0 to 72.0] | 28.9 [4.0 to 78.0] | 28.0 [4.0 to 86.7]
Pain Catastrophizing Scale - Short Form 6 (PCS-SF6) [Mean (Standard Deviation); unit: units on a scale] — A 6-item questionnaire used to assess pain-specific psychosocial construct comprising cognitive and emotional processes such as helplessness, pessimism, rumination about pain-related symptoms. The 5-point Likert scale responses are ranging from 0 (not at all) to 4 (all the time). Scores range from 0 to 24 with higher scores indicating greater pain catastrophizing.
  units on a scale | 11.6 (5.3) | 10.4 (4.5) | 10.9 (4.9) | 11.7 (5.0) | 11.1 (5.0)
Pain Detect Neuropathic Pain Questionnaire (painDETECT) Raw Score [Count of Participants; unit: Participants] — Measures the presence of neuropathic pain by summing the Likert scale responses of 'never' (0) to 'very strongly' (5) for 7-items. The total raw score ranges from 0 to 35 with higher scores indicating a worse outcome.
  Participants
    Nociceptive Pain | 136 | 154 | 142 | 147 | 579
    Possible Neuropathic Pain | 38 | 33 | 35 | 36 | 142
    Neuropathic Pain | 28 | 11 | 20 | 20 | 79
    Missing | 1 | 0 | 2 | 2 | 5
Patient Health Questionnaire-2 (PHQ-2): Raw Score [Mean (Standard Deviation); unit: units on a scale] — The PHQ-2 is a 2-item Likert-scale (0=Not at all to 3=Nearly every day) screening tool to assess depression. The score has a range of 0 to 6. A score of 3 is the optimal cut point when using the PHQ-2 to screen for depression. A higher score indicates more likely depression.
  units on a scale | 1.6 (1.6) | 1.2 (1.2) | 1.4 (1.6) | 1.6 (1.6) | 1.5 (1.5)
Healing Encounters and Attitudes Lists (HEAL) Positive Outlook: Raw Score [Mean (Standard Deviation); unit: units on a scale] — HEAL is a validated item-bank comprised of 6 domains developed through the Patient Reported Outcomes Measurement Information System (PROMIS) methodology. HEAL measures patient-reported aspects of healing encounters and attitudes. This includes evaluating factors like the patient's perception of the communication with their provider, the overall quality of care, and their feelings about the treatment process. Range for raw score was 6 to 30 and a T-score range of 21.3 to 69.3. A T-score of 50 is equal to the mean and is considered normal. Higher scores indicate more positive perception.
  units on a scale | 21.6 (5.6) | 23.0 (4.9) | 21.6 (5.8) | 21.2 (5.4) | 21.8 (5.4)
PROMIS Cognitive Function and Abilities - Short Form 2a Raw Score [Mean (Standard Deviation); unit: units on a scale] — The Patient-Reported Outcomes Measurement Information System (PROMIS) Cognitive Function and Abilities Short Form 2a assesses cognitive function and abilities. Raw scores (range 2 to 10) on the survey are converted to T scores (range 29.5 to 61.2), which are standardized scores based on the average in the population; a score of 50 would indicate meeting the average (mean) physical function T score in the reference general population, with a standard deviation of 10. Higher scores reflect greater cognitive function and abilities.
  units on a scale | 7.2 (1.8) | 7.5 (1.6) | 7.1 (1.8) | 7.2 (1.8) | 7.3 (1.8)
General Sensory Sensitivity Score (GSS) - External [Mean (Standard Deviation); unit: units on a scale] — The GSS assesses sensory sensitivity across the five external senses, as well as interoception, based on Yes (1) or No (0) responses. The GSS external score is the sum of five items with scores ranging from 0 to 5 with a higher score indicating a worse outcome.
  units on a scale | 0.9 (1.4) | 0.7 (1.2) | 1.1 (1.5) | 0.9 (1.3) | 0.9 (1.3)
General Sensory Sensitivity (GSS) Score - Interoception [Mean (Standard Deviation); unit: units on a scale] — The GSS assesses sensory sensitivity across the five external senses, as well as interoception, based on Yes (1) or No (0) responses. The GSS interoception score is the sum of three items with scores ranging from 0 to 3 with a higher score indicating a worse outcome.
  units on a scale | 0.6 (0.8) | 0.4 (0.7) | 0.6 (0.8) | 0.6 (0.8) | 0.6 (0.8)
General Sensory Sensitivity (GSS) Score - Total [Mean (Standard Deviation); unit: units on a scale] — The GSS assesses sensory sensitivity across the five external senses, as well as interoception, based on Yes (1) or No (0) responses. The total score is the sum of all 8 items with scores ranging from 0 to 8 with a higher score indicating a worse outcome.
  units on a scale | 1.5 (1.8) | 1.1 (1.6) | 1.7 (2.0) | 1.5 (1.8) | 1.5 (1.8)
Self-reported Sleep Duration in the Past Month (hours) [Mean (Standard Deviation); unit: hours] | 6.6 (1.2) | 6.7 (1.5) | 6.5 (1.2) | 6.6 (1.6) | 6.6 (1.4)
Symptom Severity Index [Mean (Standard Deviation); unit: units on a scale] — The Symptom Severity Index indicates severity of symptoms in the past week and past 6 months. The score ranges from 0 to 13 with a higher score indicating a worse outcome.
  units on a scale | 5.5 (2.9) | 4.8 (2.4) | 5.5 (2.9) | 5.9 (2.7) | 5.5 (2.8)
Widespread Pain Inventory: Raw Score [Mean (Standard Deviation); unit: units on a scale] — The Widespread Pain Inventory (WPI) measures chronic pain. The WPI score has a range 0-19. A higher score indicates more pain.
  units on a scale | 2.3 (1.8) | 2.1 (1.8) | 2.4 (1.9) | 2.5 (1.7) | 2.3 (1.8)
Stomach Pain in the Past 4 Weeks [Count of Participants; unit: Participants]
  Not bothered at all | 111 | 120 | 106 | 109 | 446
  Bothered a little | 71 | 66 | 78 | 77 | 292
  Bothered a lot | 19 | 12 | 15 | 18 | 64
  Missing | 2 | 0 | 0 | 1 | 3
Headaches in the Past 4 Weeks [Count of Participants; unit: Participants]
  Not bothered at all | 86 | 90 | 85 | 77 | 338
  Bothered a little | 95 | 96 | 92 | 103 | 386
  Bothered a lot | 20 | 12 | 22 | 24 | 78
  Missing | 2 | 0 | 0 | 1 | 3
Radiating Pain to Buttock/Thigh, Past 2 Weeks [Count of Participants; unit: Participants]
  Yes | 117 | 101 | 121 | 132 | 471
  No | 65 | 77 | 66 | 62 | 270
  Not Sure | 19 | 20 | 12 | 10 | 61
  Missing | 2 | 0 | 0 | 1 | 3
Radiating Pain to Below Knee, Past 2 Weeks [Count of Participants; unit: Participants]
  Yes | 53 | 40 | 52 | 56 | 201
  No | 126 | 143 | 136 | 132 | 537
  Not Sure | 22 | 15 | 11 | 16 | 64
  Missing | 2 | 0 | 0 | 1 | 3
Social Determinants of Health (SDOH): Transportation Needs [Count of Participants; unit: Participants] — The SDOH screening tool is a questionnaire used to assess an individual's social needs, which can impact their health. The score for transportation ranges from 0 (no) to 1 (yes) with 1 being a worse outcome.
  Participants
    Yes | 17 | 13 | 14 | 18 | 62
    No | 184 | 185 | 185 | 186 | 740
    Missing | 2 | 0 | 0 | 1 | 3
Social Determinants of Health (SDOH): Healthcare Needs [Count of Participants; unit: Participants] — The SDOH screening tool is a questionnaire used to assess an individual's social needs, which can impact their health. The score for healthcare needs ranges from 0 (no) to 1 (yes) with 1 being a worse outcome.
  Participants
    Yes | 33 | 28 | 37 | 31 | 129
    No | 168 | 170 | 162 | 173 | 673
    Missing | 2 | 0 | 0 | 1 | 3
Social Determinants of Health: Food Insecurity [Count of Participants; unit: Participants] — The SDOH screening tool is a questionnaire used to assess an individual's social needs, which can impact their health. The score for food insecurity ranges from 0 (never true) to 2 (often true) with a higher score being a worse outcome.
  Participants
    Often True | 7 | 3 | 7 | 7 | 24
    Sometimes True | 27 | 17 | 24 | 32 | 100
    Never True | 167 | 178 | 168 | 165 | 678
    Missing | 2 | 0 | 0 | 1 | 3
Social Determinants of Health (SDOH): Food Money [Count of Participants; unit: Participants] — The SDOH screening tool is a questionnaire used to assess an individual's social needs, which can impact their health. The score for food money ranges from 0 (never true) to 2 (often true) with a higher score being a worse outcome.
  Participants
    Often True | 5 | 4 | 7 | 6 | 22
    Sometimes True | 20 | 9 | 21 | 22 | 72
    Never True | 176 | 185 | 171 | 176 | 708
    Missing | 2 | 0 | 0 | 1 | 3
Social Determinants of Health (SDOH): Utilities [Count of Participants; unit: Participants] — The SDOH screening tool is a questionnaire used to assess an individual's social needs, which can impact their health. The score for health utilities ranges from 0 (no) to 1 (yes) with 1 being a worse outcome.
  Participants
    Yes | 5 | 9 | 6 | 11 | 31
    No | 196 | 189 | 193 | 193 | 771
    Missing | 2 | 0 | 0 | 1 | 3
Social Determinants of Health (SDOH): Stable Housing [Count of Participants; unit: Participants] — The SDOH screening tool is a questionnaire used to assess an individual's social needs, which can impact their health. The score for stable housing ranges from 0 (no) to 1 (yes) with 1 being a worse outcome.
  Participants
    Yes | 14 | 6 | 12 | 16 | 48
    No | 187 | 192 | 187 | 188 | 754
    Missing | 2 | 0 | 0 | 1 | 3
Social Determinants of Health (SDOH): Emotional Support [Count of Participants; unit: Participants] — The SDOH screening tool is a questionnaire used to assess an individual's social needs, which can impact their health. The score for emotional support ranges from 0 (no) to 1 (yes) with 1 being a worse outcome.
  Participants
    Yes | 185 | 180 | 184 | 187 | 736
    No | 16 | 17 | 15 | 17 | 65
    Missing | 2 | 1 | 0 | 1 | 4
Social Determinants of Health (SDOH): Number of Close Friends [Count of Participants; unit: Participants] — The SDOH screening tool is a questionnaire used to assess an individual's social needs, which can impact their health. The score for number of close friends ranges from 0-10 with a higher number indicating more friends.
  Participants
    0 | 1 | 8 | 6 | 2 | 17
    1-2 | 46 | 41 | 46 | 49 | 182
    3-5 | 99 | 89 | 90 | 94 | 372
    6-10 | 36 | 40 | 40 | 48 | 164
    More than 10 | 19 | 20 | 17 | 11 | 67
    Missing | 2 | 0 | 0 | 1 | 3
Perceived Discrimination: Race/Ethnicity [Count of Participants; unit: Participants] — Participants indicate how many times they have been treated unfairly over the course of their lives related to race/ethnicity. To score this scale, researchers add the number of events that happened at least once for the respondent. Higher scores on this scale mean more experiences of lifetime discrimination.
  Participants
    Never | 113 | 120 | 115 | 126 | 474
    Rarely | 47 | 42 | 45 | 40 | 174
    Sometimes | 40 | 36 | 39 | 38 | 153
    Often to Almost Always | 0 | 0 | 0 | 0 | 0
    Not sure | 0 | 0 | 0 | 0 | 0
    Missing | 3 | 0 | 0 | 1 | 4
Perceived Discrimination: Orientation/Gender Identity [Count of Participants; unit: Participants] — Participants indicate how many times they have been treated unfairly over the course of their lives related to orientation/gender identity. To score this scale, researchers add the number of events that happened at least once for the respondent. Higher scores on this scale mean more experiences of lifetime discrimination.
  Participants
    Never | 161 | 172 | 159 | 166 | 658
    Rarely | 24 | 16 | 20 | 19 | 79
    Sometimes | 16 | 10 | 20 | 19 | 65
    Often to Almost Always | 0 | 0 | 0 | 0 | 0
    Not sure | 0 | 0 | 0 | 0 | 0
    Missing | 2 | 0 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Patient-Reported Pain Intensity and Interference Score
Description: Patient-reported pain intensity and interference is measured by the Pain, Enjoyment of Life, and General Activity (PEG) scale. The PEG is a series of 3 questions. Results range from -10 to 10, with higher scores indicating increased pain intensity and interference at 24 Weeks compared to Baseline.
Time Frame: Baseline, 24 Weeks
Population: The analysis population is the all-randomized population to Stage 1 interventions.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stage 1: Acceptance and Commitment Therapy (ACT) | Stage 1: Duloxetine | Stage 1: Evidence Based Exercise and Manual Therapy (EBEM) | Stage 1: Enhanced Self-Care Therapy (ESC)
Number analyzed (Participants) | 203 | 198 | 199 | 205
score on a scale | 4.16 [3.74 to 4.58] | 3.86 [3.43 to 4.28] | 3.57 [3.15 to 3.99] | 4.72 [4.3 to 5.14]

2. Secondary Outcome: Patient-Reported Outcomes Measurement Information System-Pain Interference
Description: Pain interference is measured by the 4-item PROMIS (Patient-Reported Outcomes Measurement Information System) Pain Interference scale (PROMIS-PI, 4a). The PROMIS-PI, 4a is a series of 4 questions, and measures self-reported consequences of pain on relevant aspects of one's life. Results range from -34 to 34 (t-scores range from 41.6 to 75.6). For each t-score, 50 indicates the population mean with a standard deviation of 10. Lower scores indicate lower pain interference and a better outcome. PROMIS measures are not used for clinical decision making but to describe participant symptoms.
Time Frame: Baseline, 24 Weeks
Population: The analysis population is the all-randomized population to Stage 1 interventions.
Measure: Least Squares Mean (95% Confidence Interval); unit: t-scores
Arm/Group | Stage 1: Acceptance and Commitment Therapy (ACT) | Stage 1: Duloxetine | Stage 1: Evidence Based Exercise and Manual Therapy (EBEM) | Stage 1: Enhanced Self-Care Therapy (ESC)
Number analyzed (Participants) | 203 | 198 | 199 | 205
t-scores | 59.03 [57.67 to 60.39] | 58.48 [57.12 to 59.84] | 57.61 [56.25 to 58.97] | 60.13 [58.77 to 61.49]

3. Secondary Outcome: Number of Participants Self-Reporting Taking Opioids
Description: The number of participants self-reporting taking opioids ("Yes" response) is measured by a single question, "Are you currently taking any opioid pain medication on a daily basis?".
Time Frame: 24 Weeks
Population: The analysis population is the all-randomized population to Stage 1 interventions.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Acceptance and Commitment Therapy (ACT) | Stage 1: Duloxetine | Stage 1: Evidence Based Exercise and Manual Therapy (EBEM) | Stage 1: Enhanced Self-Care Therapy (ESC)
Number analyzed (Participants) | 203 | 198 | 199 | 205
Participants | 8 | 6 | 8 | 9

4. Secondary Outcome: Patient-Reported Outcomes Measurement Information System- Physical Function
Description: Physical function is measured by the Patient-Reported Outcomes Measurement Information System-Physical Function (PROMIS-PF) Short Form 6b. The PROMIS-PF Short Form 6b is a series of 6 questions. T-scores range from 21.6 to 58.7 and for each t-score, 50 indicates the population mean with a standard deviation of 10. Results range from -37.1 to 37.1, with higher physical function scores indicating a better outcome and increased physical functioning at 24 Weeks compared to Baseline. A higher physical function is the better outcome. PROMIS measures are not used for clinical decision making but to describe participant symptoms.
Time Frame: Baseline, 24 Weeks
Population: The analysis population is the all-randomized population to Stage 1 interventions.
Measure: Least Squares Mean (95% Confidence Interval); unit: t-scores
Arm/Group | Stage 1: Acceptance and Commitment Therapy (ACT) | Stage 1: Duloxetine | Stage 1: Evidence Based Exercise and Manual Therapy (EBEM) | Stage 1: Enhanced Self-Care Therapy (ESC)
Number analyzed (Participants) | 203 | 198 | 199 | 205
t-scores | 42.14 [40.81 to 43.46] | 43.32 [41.99 to 44.64] | 43.11 [41.78 to 44.43] | 41.18 [39.86 to 42.5]

5. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Depression Score
Description: Depression score is measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) 4-item depression scale from the PROMIS 29 profile. The PROMIS 4-item depression scale from the PROMIS 29 profile is a series of 4 questions. T-scores range from 41.0 to 79.4), and for each t-score, 50 indicates the population mean with a standard deviation of 10. Results range from -38.4 to 38.4, with higher scores indicating increased depression at 24 Weeks compared to Baseline. A lower depression score is the better outcome. PROMIS measures are not used for clinical decision making but to describe participant symptoms.
Time Frame: Baseline, 24 Weeks
Population: The analysis population is the all-randomized population to Stage 1 interventions.
Measure: Least Squares Mean (95% Confidence Interval); unit: t-scores
Arm/Group | Stage 1: Acceptance and Commitment Therapy (ACT) | Stage 1: Duloxetine | Stage 1: Evidence Based Exercise and Manual Therapy (EBEM) | Stage 1: Enhanced Self-Care Therapy (ESC)
Number analyzed (Participants) | 203 | 198 | 199 | 205
t-scores | 49.22 [47.71 to 50.74] | 47.83 [46.32 to 49.35] | 49.03 [47.51 to 50.54] | 50.19 [48.68 to 51.71]

6. Secondary Outcome: Patient-Reported Outcomes Measurement Information System-Emotional Distress-Anxiety
Description: Anxiety score is measured by the Patient-Reported Outcomes Measurement Information System-Emotional Distress-Anxiety (PROMIS-EDA) scale 4a. The PROMIS-EDA 4a is a series of 4 questions. T-scores range from 40.3 to 81.6, and for each t-score, 50 indicates the population mean with a standard deviation of 10. Results range from -41.3 to 41.3, with higher scores indicating increased anxiety at 24 Weeks compared to Baseline. A lower anxiety score is the better outcome. PROMIS measures are not used for clinical decision making but to describe participant symptoms.
Time Frame: Baseline, 24 Weeks
Population: The analysis population is the all-randomized population to Stage 1 interventions.
Measure: Least Squares Mean (95% Confidence Interval); unit: t-scores
Arm/Group | Stage 1: Acceptance and Commitment Therapy (ACT) | Stage 1: Duloxetine | Stage 1: Evidence Based Exercise and Manual Therapy (EBEM) | Stage 1: Enhanced Self-Care Therapy (ESC)
Number analyzed (Participants) | 203 | 198 | 199 | 205
t-scores | 49.73 [48.1 to 51.35] | 48.15 [46.52 to 49.77] | 49.14 [47.52 to 50.77] | 50.43 [48.8 to 52.05]

7. Secondary Outcome: Patient-Reported Outcomes Measurement Information System - Sleep Disturbance
Description: Sleep disturbance is measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) short form 6a. The PROMIS short form 6a is a series of 6 questions. T-scores range from 31.7 to 76.1 and for each t-score, 50 indicates the population mean with a standard deviation of 10). Results range from -44.4 to 44.4, with higher scores indicating increased sleep disturbance at 24 Weeks compared to Baseline. A lower sleep disturbance score is the better outcome. PPROMIS measures are not used for clinical decision making but to describe participant symptoms.
Time Frame: Baseline, 24 Weeks
Population: The analysis population is the all-randomized population to Stage 1 interventions.
Measure: Least Squares Mean (95% Confidence Interval); unit: t-scores
Arm/Group | Stage 1: Acceptance and Commitment Therapy (ACT) | Stage 1: Duloxetine | Stage 1: Evidence Based Exercise and Manual Therapy (EBEM) | Stage 1: Enhanced Self-Care Therapy (ESC)
Number analyzed (Participants) | 203 | 198 | 199 | 205
t-scores | 52.61 [50.98 to 54.25] | 51.45 [49.82 to 53.09] | 51.91 [50.28 to 53.54] | 53.21 [51.58 to 54.84]

8. Secondary Outcome: Sleep Duration
Description: Sleep duration is measured by the Back Pain Consortium (BACPAC) sleep duration question, "During the past month, how many hours and minutes of actual sleep did you get at night? (This may be different than the number of hours and minutes you spent in bed)." Participants respond with a number of hours and minutes. Results range from -24 to 24 hours, with higher number of hours indicating increased sleep duration at 24 Weeks compared to Baseline.
Time Frame: Baseline, 24 Weeks
Population: The analysis population is the all-randomized population to Stage 1 interventions.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Stage 1: Acceptance and Commitment Therapy (ACT) | Stage 1: Duloxetine | Stage 1: Evidence Based Exercise and Manual Therapy (EBEM) | Stage 1: Enhanced Self-Care Therapy (ESC)
Number analyzed (Participants) | 203 | 198 | 199 | 205
units on a scale | 6.82 [6.58 to 7.06] | 6.74 [6.49 to 6.98] | 6.73 [6.49 to 6.97] | 6.67 [6.43 to 6.91]

ADVERSE EVENTS:
Time Frame: All adverse events were recorded between the time the participant provided informed consent at Week -2 (Run-in Period: Weeks -2 to 0) through 4 weeks after their last treatment (Stage 1 intervention period: Weeks 0 to 12; Stage 2 intervention period: Weeks 12 to 24), up to 30 weeks.
Groups:
- Stage 2: Acceptance and Commitment Therapy (ACT): Participants newly randomized to ACT in Stage 2 will take part in 12 sessions over the course of 12 weeks. Sessions will be delivered as a combination of 4 remote face-to-face visits with a therapist and 8 therapist-supported online sessions (self-directed online modules supported by provider coaching). Participants assigned to maintain ACT will be encouraged to continue at-home skills and will have access to all previously viewed online content. In addition, participants will have access to 11 additional online ACT audio modules, but without the communications with the therapist.
- Stage 2: Duloxetine: Study participants will be treated with duloxetine for 12 weeks during the active treatment phase. All participants will be assessed at the midpoint of the intervention treatment period (Week 18) for tolerance, adverse events, and response. At the midpoint phone call:
  Participants tolerating the medication with no side effects will be instructed to increase to 60mg/day (if currently taking 30mg/day) or remain on their current dosage (if currently taking 60mg/day).
- Stage 2: Evidence Based Exercise and Manual Therapy (EBEM): Participants newly randomized to EBEM in stage 2 will take part in a total of 10 sessions over an 8-week treatment period. Two sessions per week are provided in the first two weeks followed by weekly sessions over the next 6 weeks. Treatment sessions will last approximately 60 minutes each. Participants assigned to maintain EBEM will receive 4 additional in-person EBEM sessions during weeks 1-4 of this period. If visits are missed and/or need to be rescheduled, visits may be scheduled up to 5 weeks from the date of the first augmenting/maintenance visit.
- Stage 2: Enhanced Self-Care Therapy (ESC): Participants newly randomized to ESC in stage 2 will be provided modules digitally for self-administration over a period of 12 weeks. There will be no therapist associated with the delivery of these educational materials; however, after the first four modules, email or text messages will be used to make personalized recommendations for accessing additional modules based upon identified problems from the baseline assessment. Additionally, the walking program module will utilize Fitbit step tracking to allow participants to monitor their walking progress. Participants assigned to maintain ESC in the second period intervention will receive personalized recommendations based on the most recently completed PROMIS 29+2.
- Stage 2: ACT and Duloxetine: Participants received both ACT and duloxetine in Stage 2. Participants who received augmented Stage 2 treatments always continued their stage 1 treatment. The continued intervention matches the dose of those maintaining Stage 1 treatment alone, and the added intervention is as if they were newly randomized.
- Stage 2: ACT and EBEM: Participants received both ACT and EBEM in Stage 2. Participants who received augmented Stage 2 treatments always continued their stage 1 treatment. The continued intervention matches the dose of those maintaining Stage 1 treatment alone, and the added intervention is as if they were newly randomized.
- Stage 2: ACT and ESC: Participants received both ACT and ESC in Stage 2. Participants who received augmented Stage 2 treatments always continued their stage 1 treatment. The continued intervention matches the dose of those maintaining Stage 1 treatment alone, and the added intervention is as if they were newly randomized.
- Stage 2: Duloxetine and EBEM: Participants received both duloxetine and EBEM in Stage 2. Participants who received augmented Stage 2 treatments always continued their stage 1 treatment. The continued intervention matches the dose of those maintaining Stage 1 treatment alone, and the added intervention is as if they were newly randomized.
- Stage 2: Duloxetine and ESC: Participants received both duloxetine and ESC in Stage 2. Participants who received augmented Stage 2 treatments always continued their stage 1 treatment. The continued intervention matches the dose of those maintaining Stage 1 treatment alone, and the added intervention is as if they were newly randomized.
- Stage 2: EBEM and ESC: Participants received both EBEM and ESC in Stage 2. Participants who received augmented Stage 2 treatments always continued their stage 1 treatment. The continued intervention matches the dose of those maintaining Stage 1 treatment alone, and the added intervention is as if they were newly randomized.
Arm/Group | Stage 1: Acceptance and Commitment Therapy (ACT) | Stage 1: Duloxetine | Stage 1: Evidence Based Exercise and Manual Therapy (EBEM) | Stage 1: Enhanced Self-Care Therapy (ESC) | Stage 2: Acceptance and Commitment Therapy (ACT) | Stage 2: Duloxetine | Stage 2: Evidence Based Exercise and Manual Therapy (EBEM) | Stage 2: Enhanced Self-Care Therapy (ESC) | Stage 2: ACT and Duloxetine | Stage 2: ACT and EBEM | Stage 2: ACT and ESC | Stage 2: Duloxetine and EBEM | Stage 2: Duloxetine and ESC | Stage 2: EBEM and ESC
All-Cause Mortality (participants affected / at risk) | 0/191 | 0/172 | 0/184 | 0/205 | 0/65 | 0/71 | 0/110 | 0/85 | 0/33 | 0/52 | 0/84 | 0/22 | 0/54 | 0/85
Serious Adverse Events (participants affected / at risk) | 4/191 | 1/172 | 6/184 | 2/205 | 4/65 | 0/71 | 3/110 | 2/85 | 1/33 | 0/52 | 4/84 | 0/22 | 1/54 | 4/85
Other Adverse Events (participants affected / at risk) | 2/191 | 92/172 | 7/184 | 4/205 | 1/65 | 29/71 | 3/110 | 0/85 | 12/33 | 3/52 | 2/84 | 4/22 | 18/54 | 5/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1: Acceptance and Commitment Therapy (ACT) (N=191) | Stage 1: Duloxetine (N=172) | Stage 1: Evidence Based Exercise and Manual Therapy (EBEM) (N=184) | Stage 1: Enhanced Self-Care Therapy (ESC) (N=205) | Stage 2: Acceptance and Commitment Therapy (ACT) (N=65) | Stage 2: Duloxetine (N=71) | Stage 2: Evidence Based Exercise and Manual Therapy (EBEM) (N=110) | Stage 2: Enhanced Self-Care Therapy (ESC) (N=85) | Stage 2: ACT and Duloxetine (N=33) | Stage 2: ACT and EBEM (N=52) | Stage 2: ACT and ESC (N=84) | Stage 2: Duloxetine and EBEM (N=22) | Stage 2: Duloxetine and ESC (N=54) | Stage 2: EBEM and ESC (N=85)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulcer (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cat scratch disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Magnetic resonance imaging abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testis cancer (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Physical assault (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychiatric care (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1: Acceptance and Commitment Therapy (ACT) (N=191) | Stage 1: Duloxetine (N=172) | Stage 1: Evidence Based Exercise and Manual Therapy (EBEM) (N=184) | Stage 1: Enhanced Self-Care Therapy (ESC) (N=205) | Stage 2: Acceptance and Commitment Therapy (ACT) (N=65) | Stage 2: Duloxetine (N=71) | Stage 2: Evidence Based Exercise and Manual Therapy (EBEM) (N=110) | Stage 2: Enhanced Self-Care Therapy (ESC) (N=85) | Stage 2: ACT and Duloxetine (N=33) | Stage 2: ACT and EBEM (N=52) | Stage 2: ACT and ESC (N=84) | Stage 2: Duloxetine and EBEM (N=22) | Stage 2: Duloxetine and ESC (N=54) | Stage 2: EBEM and ESC (N=85)
Constipation (Gastrointestinal disorders) | 0 (0) | 17 (18) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 33 (34) | 0 (0) | 0 (0) | 0 (0) | 14 (14) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 2 (2) | 9 (9) | 0 (0)
Fatigue (General disorders) | 0 (0) | 21 (21) | 2 (2) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 1 (1)
Irritability (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 12 (12) | 1 (1) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 0 (0)
Insomnia (Nervous system disorders) | 0 (0) | 11 (11) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 16 (17) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Vascular disorders) | 0 (0) | 12 (12) | 0 (0) | 2 (2) | 0 (0) | 8 (8) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
The BEST Trial is a sequential, multiple-assignment randomized trial designed to estimate the optimal treatment (or sequence) for chronic low back pain based on unique biomarkers and response to treatment. As this precision-medicine focus dictates individualized rather than arm-level contrasts, no between-arm comparative-effectiveness analyses are planned as primary analyses. The primary goal of this study was to identify predictive biomarkers for each treatment not comparative effectiveness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT05396014/Prot_001.pdf
  • Statistical Analysis Plan (2025-05-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT05396014/SAP_002.pdf
  • Informed Consent Form (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/14/NCT05396014/ICF_000.pdf